CLINICAL TRIAL: NCT00420472
Title: An Open-Label Study to Evaluate the Effect on Quality of Life of Switching Kidney Transplant Patients From Reduced Dose EC-MPS to a Higher Than the Equimolar Dose of CellCept
Brief Title: A Study of CellCept (Mycophenolate Mofetil) in Kidney Transplant Patients Switched From EC-MPS.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20240
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: mycophenolate mofetil [CellCept]

SUMMARY:
This study will assess the safety, efficacy and effect on quality of life of switching kidney transplant patients from reduced dose EC-MPS treatment due to gastrointestinal problems to a higher than the equimolar dose of CellCept. Patients will be switched, initially, from EC-MPS (<1440g/day) to an equimolar dose of CellCept, and at the next visit (day 10 +/- 5) the CellCept dose will be increased by 250mg/day, and the daily dose will be split into 3-4 doses. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* first or second kidney transplant;
* EC-MPS therapy for >=6 months, with a stable dose for >=2 months;
* lower than recommended dose of EC-MPS (<1440g/day) due to gastrointestinal complaints.

Exclusion Criteria:

* patients who have participated in this study before;
* patients currently participating in another clinical trial, or who participated in one during the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-03

PRIMARY OUTCOMES:
Gastrointestinal Quality of Life index, and Gastrointestinal Symptom Rating Scale, at 3 months.

SECONDARY OUTCOMES:
Efficacy: Mean dose increase of CellCept. Pharmacokinetics: Comparison of pharmacokinetic parameters under EC-MPS and CellCept therapy. Safety: AEs; acute rejection episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Germany (6):
  - Berlin
  - Cologne
  - Dresden
  - Essen
  - Hanover
  - Münster